CLINICAL TRIAL: NCT04929119
Title: The Effect of Wearing Orthokeratology on Objective Visual Quality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: XiaoYong Liu (Other)
Responsible Party: Sponsor-Investigator, XiaoYong Liu, Deputy chief physician, First Affiliated Hospital of Jinan University
Organization: First Affiliated Hospital of Jinan University (Other)
Other Study IDs: 2021jnU
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Visual Quality
Keywords: Objective visual quality; Orthokeratology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Before wearing the Orthokeratology: OPD-Scan was performed and the following data were recorded: 4 mm high order strehl ratio (SR) , 4 mm high order corneal aberrations (Hoa ) , Spherical Aberrations (SA) , Coma Aberrations (Coma) , Trefoil Aberrations (RMS) , corneal aspheric index (Q, e) , corneal surface regularity index (SRI) , corneal surface asymmetry index (Sai)
- Wear Orthokeratology for a week: OPD-Scan was performed and the following data were recorded: 4 mm high order strehl ratio (SR) , 4 mm high order corneal aberrations (Hoa ) , Spherical Aberrations (SA) , Coma Aberrations (Coma) , Trefoil Aberrations (RMS) , corneal aspheric index (Q, e) , corneal surface regularity index (SRI) , corneal surface asymmetry index (Sai)
- Wear Orthokeratology for a month: OPD-Scan was performed and the following data were recorded: 4 mm high order strehl ratio (SR) , 4 mm high order corneal aberrations (Hoa ) , Spherical Aberrations (SA) , Coma Aberrations (Coma) , Trefoil Aberrations (RMS) , corneal aspheric index (Q, e) , corneal surface regularity index (SRI) , corneal surface asymmetry index (Sai)
- Wear Orthokeratology for three months: OPD-Scan was performed and the following data were recorded: 4 mm high order strehl ratio (SR) , 4 mm high order corneal aberrations (Hoa ) , Spherical Aberrations (SA) , Coma Aberrations (Coma) , Trefoil Aberrations (RMS) , corneal aspheric index (Q, e) , corneal surface regularity index (SRI) , corneal surface asymmetry index (Sai)
- Wear Orthokeratology for six months: OPD-Scan was performed and the following data were recorded: 4 mm high order strehl ratio (SR) , 4 mm high order corneal aberrations (Hoa ) , Spherical Aberrations (SA) , Coma Aberrations (Coma) , Trefoil Aberrations (RMS) , corneal aspheric index (Q, e) , corneal surface regularity index (SRI) , corneal surface asymmetry index (Sai)

SUMMARY:
The visual quality indexes of these patients before and after Orthokeratology treatment were compared: 4 mm higher strehl ratio (SR) , 4 mm higher order corneal aberrations (Hoa ) , Spherical Aberrations (SA) , Comas, Trefoil Aberrations (RMS) , corneal aspheric index (Q, e) , corneal surface regularity index (SRI) , corneal surface asymmetry index (Sai)

DETAILED DESCRIPTION:
USING OPD-SCAN III instrument method: Drag The joystick to focus on the screen prompt, and the device automatically starts to measure the aberration when the yellow focus is shown; Simk will change from black to rose red when the aberration is measured to start measuring the corneal topography, prompting the patient to blink the tear film evenly and press the button on the joystick when the focus is completed.The following data were obtained and analyzed: 4 mm high order STREHL rate (SR) , 4 mm high order corneal aberration (Hoa ) , Spherical Aberration (SA) , Coma Aberration (Coma) , Trefoil Aberration (RMS) , corneal aspheric index (Q, e) , corneal surface regularity index (SRI) , corneal surface asymmetry index (Sai)

ELIGIBILITY:
Inclusion Criteria:

* The subject understands the purpose of this clinical trial and is willing, able and committed to return to the center for all clinical trial visits and to complete all research related procedures

Exclusion Criteria:

* 1. Associated with corneal abnormalities, such as active Keratitis (corneal infection) , corneal dystrophy, Keratoconus, corneal Leukoplakia, corneal hypoesthesia, or previous corneal surgery, or a history of corneal trauma;
* 2, there are other eye diseases, such as Dacryocystitis, dry eye disease, conjunctivitis, blepharitis, Uveitis, and other inflammation, Glaucoma, cataracts, fundus disease, eye tumors, ocular trauma, squint patients;
* 3. A history of allergy to contact lens or contact Lens Solution.
* 4. Test results indicate that subjects with contraindications or unsuitable for wearing Orthokeratology.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Before wearing the Orthokeratology:30cases;Wear Orthokeratology for a week:30cases;Wear Orthokeratology for a month:30cases;Wear Orthokeratology for three months:30cases;Wear Orthokeratology for six months:30cases
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-03-07 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
4 mm high-order strehl ratio | 6 months
  Objective visual quality 1
4 mm high-order corneal aberrations (Hoa) in Microns | 6 months
  Objective visual quality 2
Spherical Aberrations (SA) in Microns | 6 months
  Objective visual quality 3
Coma Aberrations (COMA) in Microns | 6 months
  Objective visual quality 4
Trefoil Aberrations in Microns | 6 months
  Objective visual quality 5
corneal aspheric index(Q) | 6 months
  Objective visual quality 6
corneal aspheric index(e) | 6 months
  Objective visual quality 7
corneal surface regularity index (SRI) | 6 months
  Objective visual quality 8
corneal surface asymmetry index (Sai) | 6 months
  Objective visual quality 9

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Jinan University, Guangdong, Guangzhou, China

REFERENCES:
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Background] Swarbrick HA. Orthokeratology review and update. Clin Exp Optom. 2006 May;89(3):124-43. doi: 10.1111/j.1444-0938.2006.00044.x. PMID 16637967
- [Background] Goldstone RN, Yildiz EH, Fan VC, Asbell PA. Changes in higher order wavefront aberrations after contact lens corneal refractive therapy and LASIK surgery. J Refract Surg. 2010 May;26(5):348-55. doi: 10.3928/1081597X-20100218-03. Epub 2010 May 19. PMID 20506992
- [Background] Yin Y, Zhao Y, Wu X, Jiang M, Xia X, Chen Y, Song W, Hu S, Zhou X, Young K, Wen D. One-year effect of wearing orthokeratology lenses on the visual quality of juvenile myopia: a retrospective study. PeerJ. 2019 May 30;7:e6998. doi: 10.7717/peerj.6998. eCollection 2019. PMID 31179186
- [Background] Lian Y, Shen M, Huang S, Yuan Y, Wang Y, Zhu D, Jiang J, Mao X, Wang J, Lu F. Corneal reshaping and wavefront aberrations during overnight orthokeratology. Eye Contact Lens. 2014 May;40(3):161-8. doi: 10.1097/ICL.0000000000000031. PMID 24681612
- [Derived] Cheng Z, Meng J, Ye L, Wang X, Gong Y, Liu X. Changes in the Objective Vision Quality of Adolescents in a Mesopic Visual Environment After Wearing Orthokeratology Lenses: A Prospective Study. Eye Contact Lens. 2024 Sep 1;50(9):384-394. doi: 10.1097/ICL.0000000000001111. Epub 2024 Jul 3. PMID 38968599